CLINICAL TRIAL: NCT07282119
Title: Can EmeraldLED Reshape Your Body With Continued Use?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 44804
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Body Composition

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single Arm observational where participants act as their own control
  Interventions: Device: EmeraldLED

INTERVENTIONS:
Device: EmeraldLED — This device is a customizable, multi-wavelength therapeutic system designed for individualized cosmetic treatments. It features an easy-to-use interface with preprogrammed treatment categories, a wide pulsing frequency range from 1 to 15,000 Hz, and independent wavelength control for precise protocol tailoring. The system delivers five wavelengths-450 nm, 525 nm, 650 nm, 810 nm, and 980 nm-with an output power of 3,325 W and irradiance up to 119 mW/cm².
  The green light EmeraldLED therapy provided in this study is set at 525 nm.

SUMMARY:
Already using EmeraldLED? TheGreen Light Therapy study explores how continuing participants' 15-minute sessions, twice a week, may continue to support positive changes in body composition.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to rigorously explore the efficacy of green light therapy on body composition and overall well-being, under the leadership of Ryan, the CEO of beem® Light Sauna. With over 30 years of experience in the wellness industry, Ryan has observed firsthand the surge in popularity of green light therapy, accompanied by a myriad of claims regarding its benefits. Despite widespread anecdotal evidence suggesting that green light therapy can aid in weight loss and improve mood, there remains a significant gap in scientific research to support these claims conclusively. This study aims to bridge this gap by providing empirical evidence on the effects of green light therapy.

The objective of this study is to empower participants with knowledge about how green light exposure might influence their weight management efforts and overall sense of well-being. By participating in this remote trial, individuals will receive personalized data regarding changes in their body composition and mood, following a structured regimen of green light therapy. This personalized feedback will enable participants to make informed decisions about incorporating green light therapy into their health and wellness routines.

The significance of this study lies in its potential to challenge and possibly redefine existing weight management strategies. By collecting and analyzing data on how green light therapy affects individuals, this study seeks to provide insights that could lead to new, innovative approaches to health and wellness. While acknowledging the limitations of this initial trial, including the necessity for further comprehensive research, the findings could serve as a valuable foundation for future studies and health innovations.

In sum, this decentralized trial represents a critical step towards demystifying the effects of green light therapy on body composition and mood enhancement. Through rigorous scientific investigation, this study aims to validate or debunk the claims surrounding green light therapy, thereby contributing to the broader understanding of its potential benefits and limitations. Participants' involvement is not just a journey towards personal health enlightenment but also a contribution to the global conversation on effective, science-backed wellness strategies.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with eye conditions
* Individuals not active with EmeraldLED

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Body Composition Measurement Form | Change from baseline (Day 1-3) in body measurements at 4 weeks after the start of the intervention (Day 27-33).
  The Body Composition Measurement Form is specifically crafted to accurately track changes in body measurements relevant to individuals engaged in weight loss or bodybuilding. This form allows for the consistent recording of key physical metrics across various body parts, facilitating the evaluation of fitness progress. By using this form, individuals can obtain a clear picture of the physical changes resulting from their exercise routines and nutritional choices. Each measurement is to be recorded in centimeters to maintain uniformity and precision.
Quality of Life and Health Survey | Change from baseline (Day 1-3) in quality of life and health perceptions at 4 weeks after the start of the intervention (Day 27-33).
  This survey asks about your feelings towards your quality of life, health, and various areas of your life. It covers your experiences and feelings in the past four weeks. Please choose the answer that appears most appropriate.
Body Image and Self-Perception Survey | Change from baseline (Day 1-3) in body image and self-perception at 4 weeks after the start of the intervention (Day 27-33).
  This survey aims to understand an individual's perception of their body, attractiveness, and physical functionality. It contains multiple-choice questions with five options ranging from 'Strongly Disagree' to 'Strongly Agree'. The questions are divided into three categories: Body Satisfaction, Attractiveness Evaluation, and Physical Functionality Awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=44799